CLINICAL TRIAL: NCT00658489
Title: Implementation and Evaluation of Bright Futures Curriculum Within CORNET Continuity Practice
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Christiana Care Health Services (Other)
Collaborators: HRSA/Maternal and Child Health Bureau (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 27092; DDD#504887
Record Dates: First submitted 2008-04-11; First posted 2008-04-15 (Estimated); Last update posted 2011-11-11 (Estimated); Status verified 2011-11

CONDITIONS: Dental Health; Iron Deficiency
MeSH Terms: conditions — Iron Deficiencies | interventions — Educational Status

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): Residents randomized to the promotion of oral health group will receive training consisting of 7 modules (3 on the Bright Futures curriculum and 4 on oral health promotion). They will then enroll 3 patient-child dyads from their practice who present for a well child care visit. Outcomes will be obtained by completing pre- and post-study surveys. Residents will be observed by a faculty preceptor during 3 different patient encounters, and will receive feedback at the end of the 6 month study period.
  Interventions: Behavioral: Education
- 2 (Active Comparator): Residents randomized to the prevention of iron deficiency group will complete one web-based module.
  Interventions: Behavioral: Education

INTERVENTIONS:
Behavioral: Education — One group of residents will receive extensive web-based training in the promotion of oral health. The second group of residents will complete a single training module in the prevention of iron deficiency. The third arm consists of parent-child dyads, who will participate in one well-child care visit.

SUMMARY:
The purpose of "Bright Futures" is to promote and improve infant, child, and adolescent health within the context of family and community. CORNET (COntinuity Research NETwork of the Ambulatory Pediatric Association) is a national practice-based research network of resident continuity practices, whose mission is to establish a self-sustaining collaborative research network among pediatric continuing clinic clinicians who will produce quality research in primary care, health care delivery, and education.

DETAILED DESCRIPTION:
"Bright Futures" offers a child and family-centered approach to health promotion in incorporating partnership and communication skills of providers. Two areas of importance are promotion of oral health and prevention of iron deficiency. Residents will be randomized to one of these two groups and will receive web-based education about that particular topic. Residents randomized to group 1 will receive training consisting of 7 modules: 3 on the Bright Futures concepts and 4 on oral health promotion. They will be trained in performing an oral health assessment, identifying caries, and encouraged to establish a dental home for patients. They must communicate with at least one dental practice in the community to determine barriers to care, issues regarding insurance, potential solutions to improve referral, and access to dental care. Residents in group 2 will complete a single educational module on the identification and prevention of iron deficiency. They will be trained to identify iron deficiency and iron deficiency anemia, understand risk prevention strategies, improved methods of identification, and treatment.

Each resident will recruit 3 patients, children between the ages of 12-35 months, for whom he/she is the primary care provider. Each parent-child dyad will participate in one well-child care visit. Each visit will be observed by a faculty preceptor.

This study design was chosen to compare a more sophisticated and time-intensive curriculum to a more modest one. By having a curriculum with minimal overlap between the two groups, the investigators hope to examine the knowledge obtained by the residents, which health promotion aspects they address during their encounters, and to compare the establishment of a dental home in the two groups of patients.

ELIGIBILITY:
Inclusion Criteria:

* Children ages 12-35 months

Exclusion Criteria:

* None

Ages: 12 Months to 35 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 10 (Actual)
Dates: Start 2008-01; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
Residents will receive the direct benefit of exposure to a new curriculum and feedback on performance by their preceptor. Parents will benefit from greater access to their primary care providers. | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Shirley Klein, MD, Principal Investigator — Christiana Care Health Services